CLINICAL TRIAL: NCT06775171
Title: The Impact of Video-Based Pressure Injury Training on Caregivers' Knowledge Levels, Caregiving Attitudes, Behaviors, and Reactions
Brief Title: Impact of Video-Based Pressure Injury Training on Caregivers' Knowledge, Attitudes, Behaviors & Reactions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi Baran CAMCI (Other)
Responsible Party: Sponsor-Investigator, Gazi Baran CAMCI, Research Assistant, Kahramanmaraş İstiklal University
Organization: Kahramanmaraş İstiklal University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kahramanmaras Istıklal Unıv
Record Dates: First submitted 2024-08-29; First posted 2025-01-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pressure Injury
Keywords: Caregiver; Caregiving Behavior; Caregiving Response; Caregiving Attitude; Pressure Injury; Video Training
MeSH Terms: conditions — Pressure Ulcer | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- video training group (Experimental): Caregiving knowledge, attitudes, behaviors and caregiving reactions will be measured in the pre-test. Then, the participants will be given training cards containing the QR codes of the videos previously created by the researcher, they will be asked to watch them at least three times at any time and environment they want for four weeks, and weekly feedback will be received. As a post-test, knowledge level, attitude, behavior and caregiving reactions will be measured at the end of the fourth week.
  Interventions: Behavioral: video training group
- standard education group (Experimental): Caregiving knowledge, attitudes, behaviors and caregiving reactions will be measured in the pre-test. Afterwards, a verbal training will be given for twenty minutes using the training booklet prepared by the researcher in advance for the prevention of caregiving. As a post-test, knowledge, attitude, behavior and caregiving reactions will be measured face-to-face at the end of the fourth week.
  Interventions: Behavioral: video training group
- control group (No Intervention): The control group will not receive any training and measurements will be made simultaneously with the experimental groups. In the pre-test, caregiving knowledge level, attitude, behavior and caregiving reactions will be measured. As a post-test, knowledge level, attitude, behavior and caregiving reactions will be measured face to face at the end of the fourth week.

INTERVENTIONS:
Behavioral: video training group — Creation of the Education Booklet While creating the education booklet that includes the definition of BY, the areas where it frequently develops, risk factors, classification, prevention and situations where it requires professional support, it will be created by the researcher by scanning the current literature and taking the opinions of the Faculty Members from the Nursing Fundamentals field in terms of scope, comprehensibility and scientific content.
  Creation of Videos The videos will be prepared in five separate videos that will include the definition of BY, the areas where it frequently develops, risk factors, classification, prevention and situations where it requires professional support in line with the education booklet. QR codes of the prepared videos will be created. Each video will be planned to be 5-10 minutes. The videos will be checked by the Advisor Faculty Member and corrections will be made in line with his/her suggestions.
  Other Names: standard education group; control group
  Arms: standard education group; video training group

SUMMARY:
It is known that caregivers of patients at high risk of developing pressure injury (PBI) have important responsibilities and education to be given to caregivers is necessary for the prevention of PBI. This study was planned to determine the effect of video-assisted training to be given to caregivers of patients at high risk of developing BP on caregivers' knowledge level, attitudes, behaviors and reactions towards caregiving. The research will be conducted as a randomized controlled experimental study in Gaziantep City Hospital inpatient units between 15.09.2023-15.09.2025. A total of 270 patients will be included in the study, with 90 patients assigned to each of the video training group, standard training group and control group. Criterion sampling method will be used to assign the participants to the experimental and control groups, and those with medium and high Braden Pressure Ulcer Risk Assessment Scale scores will be determined and randomly assigned to the groups. Sociodemographic Characteristics Form, Braden Pressure Ulcer Risk Assessment Scale, Family Caregivers' Knowledge, Attitude and Practice Assessment Tool for Pressure Injury Prevention and Caregiver Reaction Assessment Scale will be used for data collection. Data will be collected by face-to-face interviews in inpatient units after randomization. Participants in the video training group will be shown training videos on prevention of SCI, while the standard training group will receive a verbal training and the control group will follow routine clinical protocols. They will be asked to watch the video trainings at least three times in any time and environment they want for four weeks and their weekly feedback will be collected. Final measurements of all participants will be made at the end of the fourth week. In the statistical analysis of the data, descriptive statistics, t test, ANOVA, ANCOVA, Mann Withney U, Kruskall Wallis H test and Wilcoxon signed-rank test will be used according to normal distribution.

DETAILED DESCRIPTION:
Pressure injuries (PI) are defined as localized damage to the skin and subcutaneous tissues due to pressure or shear accompanying pressure. This damage is seen in bone protrusions or in body areas that are in contact with medical devices and other objects. The main factor in the formation of PI is the decrease in blood flow to the tissues due to continuous pressure exposure. Pressure on the tissue prevents capillary circulation. As a result, capillary perfusion is impaired, adequate oxygenation of the tissues cannot be provided, and tissue ischemia develops. In cases where capillary circulation is completely blocked, PI can occur in an average of 2-6 hours. The decrease in tissue tolerance due to external factors such as friction, shear, and humidity and/or internal factors related to the patient also increases the risk of PI. PI developing in patients is known to cause physical and psychological trauma, negatively affect daily life activities, prolong the duration of hospital stay, reduce the quality of life, and increase care expenses. In Canada, the cost of BY care and treatment is determined to be between $2,450-12,648 per case, depending on the complications and stage of the injury. It has been reported that the annual cost of BY to the American healthcare system is $9.1-11.6 billion. In a systematic review conducted by Demarré et al. (2015) where 17 studies were analyzed, it was seen that the cost of treatment for BY for each patient varied between €1.7-470.5 per day, and the daily cost for preventing BY was between €2.6-87.6 per patient. In the studies, the general prevalence of BY was found to be 10.8% in European countries, 7.9% in Australia, 26% in Canada, and 15% in the United States. In a point prevalence study conducted by the Wound Ostomy Incontinence Nurses Association (YOİHD) in Turkey (2019) and covering patients from 13 hospitals in 12 regions of Turkey (n=5,088), the overall prevalence of BY was found to be 9.5%. In a study conducted with patients receiving home care services (n=2,779), the prevalence of BY was found to be 6.8% and 26.8% of patients were at risk of BY. In Australia, the prevalence of BY in the community was reported to be 9.4%, and in England, it was reported to be between 11% and 13%. In a study conducted in Turkey, the incidence of pressure ulcers in bedridden patients was determined to be 28.4%. In a study conducted with patients receiving home care services from a training and research hospital in Turkey (n=786), the BY rate was determined to be 29.8%. BY is seen as an important risk affecting the health of patients by health institutions in the world and in our country. Preventive practices are gaining importance due to the negative consequences of BY. The scope of education, which is considered an important component in the prevention of pressure injuries, should not be limited to the education of nurses only; risk factors should be taught to patients and their relatives who provide care, and training should be provided to reduce the risk. Since studies examining the effect of education on the prevention of BY do not provide sufficient evidence, more research is needed. The care process of patients with BY is made difficult due to the inability of caregivers to access educational opportunities. Inclusion of caregivers in the care team is effective in ensuring continuity of care, coordination, and the success of individual-centered BY prevention plans. In this context, in addition to training nurses, training of caregivers is important in the implementation of BY prevention plans and ensuring compliance with these plans. Training techniques for the prevention of BY include various techniques such as video-supported education, web-based education, distance education, education through tele-nursing, and standard (verbal) education. Health education includes various technologies such as collaborative applications provided through information and communication technologies and tools that enable individual learning. Educational videos, which are among these technologies, are tools that support knowledge, critical awareness and health promotion. Educational videos have been used in a number of pedagogical experiences that demonstrate the importance of their applicability in learning and teaching and combine elements such as images, sound and text under one roof. Video-assisted education is a very important technique because it concretizes what is conveyed with auditory and visual data, easily conveys scenarios related to real life and appeals to more than one sense. It is known that the use of video technology positively affects the knowledge levels of caregivers of patients with BD. Individuals who provide informal care to patients are usually family members and assume serious responsibilities. Caregivers' reactions to caregiving, in other words, the problems they experience while providing care, can also be classified as physical, social, economic and psychological problems.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Agreeing to participate in the study,
* Being literate,
* Being able to communicate verbally,
* Having a device (tablet, smartphone or computer) that can watch videos,
* Being able to provide care to a patient with a moderate or high Braden Pressure Ulcer Risk Assessment Scale score.

Exclusion Criteria:

Exclusion criteria from the study

* Refusing to participate in the study,
* Providing care to a patient with a low Braden Pressure Ulcer Risk Assessment Scale score.
* Not watching all of the videos,
* Not completing the four-week training period,
* Requesting to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 270 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Caregiver Knowledge Level | a mounth
  Changes in caregiver knowledge about pressure injuries following the video-assisted training.

SECONDARY OUTCOMES:
Attitudes Towards Caregiving-Caregiver Behaviors-Caregiver Responses | a mounth
  Changes in caregiver attitudes towards preventing pressure injuries following the training--Changes in caregiver practices towards preventing pressure injuries following the training-Changes in caregiver emotional and behavioral responses during the caregiving process following the training.

OTHER OUTCOMES:
Braden Pressure Ulcer Risk Assessment Scale Score-Video Viewing Frequency and Feedback | a mounth
  Caregiver effectiveness in risk assessment and how this score changed following the training-Analysis of the number of times they watched the video training and the feedback they received.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş İstiklal Üniversitesi, Kahramanmaraş, Oniksubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No